CLINICAL TRIAL: NCT05061589
Title: Incidence and Risk Factors of Parastomal Hernia in Patients With Permanent Colostomy in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Other Study IDs: BFH-IRFPH
Record Dates: First submitted 2021-09-20; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Hernia; Stoma Colostomy
MeSH Terms: conditions — Hernia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: permanent colostomy — An operation that creates an opening for the colon through the abdomen

SUMMARY:
Parastomal hernia refers to the protrusion of the area around the stoma or the ectopic protrusion of abdominal contents from the stoma (colostomy, ileostomy, ileostomy for bladder) in the abdominal wall defect. Parastomal hernia is one of the common complications after permanent colostomy. According to guidelines published by the European Hernia Society, the overall incidence of parastomal hernia is unknown, but it can be predicted to be over 30% at 12 months, over 40% at 2 years, and over 50% at longer follow-up periods. Parastomal hernia may have no obvious symptoms at the beginning or only protrusion around the stoma. However, with the progression of the disease, the protrusion site may gradually increase, resulting in leakage, skin ulcers, perforation, incarceration, obstruction, strangulation and other serious complications. It will seriously affect the quality of life of patients and increase the medical burden and cost.

Risk factors related to parastomal hernia are currently considered to be mainly related to the patient's own factors and surgical factors. Studies have shown that female, old age, obesity, cardiopulmonary diseases, diabetes, long-term use of cortisol and other factors can increase the incidence of parastomal hernia in patients . Methods of stoma including extraperitoneal stoma, appropriate aperture of stoma and preventive mesh placement can reduce the incidence of parastomal hernia in patients.

In this study, patients with permanent colostomy and relevant information of surgery as well as the current incidence of parastomal hernia will be retrospectively collected in some high-level and high-volume tertiary hospitals in China. This study will be helpful to provide data reference for subsequent studies in this field.

ELIGIBILITY:
Inclusion Criteria:

* permanent colostomy after colorectal surgery for benign or malignant diseases
* No previous colostomy history

Exclusion Criteria:

* No CT scan follow-up at 1 year after surgery
* Another ileocolonic diversion was performed except for the cause of parastomal hernia

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients underwent permanent colostomy after colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 712 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of parastomal hernia | 1 year after permanent colostomy

SECONDARY OUTCOMES:
Incidence of parastomal hernia | 2 year after permanent colostomy
Incidence of parastomal hernia | 5 year after permanent colostomy
risk factors of parastomal hernia | 1 year after permanent colostomy
classification of parastomal hernia | 1 year after permanent colostomy

CONTACTS AND LOCATIONS:
Overall Officials: Zhongtao Zhang, Study Chair — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University
Locations (2):
- China (2):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Beijing Friendship Hospital, Capital medical University, Beijing, Xicheng Dis

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antoniou SA, Agresta F, Garcia Alamino JM, Berger D, Berrevoet F, Brandsma HT, Bury K, Conze J, Cuccurullo D, Dietz UA, Fortelny RH, Frei-Lanter C, Hansson B, Helgstrand F, Hotouras A, Janes A, Kroese LF, Lambrecht JR, Kyle-Leinhase I, Lopez-Cano M, Maggiori L, Mandala V, Miserez M, Montgomery A, Morales-Conde S, Prudhomme M, Rautio T, Smart N, Smietanski M, Szczepkowski M, Stabilini C, Muysoms FE. European Hernia Society guidelines on prevention and treatment of parastomal hernias. Hernia. 2018 Feb;22(1):183-198. doi: 10.1007/s10029-017-1697-5. Epub 2017 Nov 13. PMID 29134456
- [Background] Hong SY, Oh SY, Lee JH, Kim DY, Suh KW. Risk factors for parastomal hernia: based on radiological definition. J Korean Surg Soc. 2013 Jan;84(1):43-7. doi: 10.4174/jkss.2013.84.1.43. Epub 2012 Dec 26. PMID 23323235
- [Background] Lian L, Wu XR, He XS, Zou YF, Wu XJ, Lan P, Wang JP. Extraperitoneal vs. intraperitoneal route for permanent colostomy: a meta-analysis of 1,071 patients. Int J Colorectal Dis. 2012 Jan;27(1):59-64. doi: 10.1007/s00384-011-1293-6. Epub 2011 Sep 3. PMID 21892608
- [Background] Pilgrim CH, McIntyre R, Bailey M. Prospective audit of parastomal hernia: prevalence and associated comorbidities. Dis Colon Rectum. 2010 Jan;53(1):71-6. doi: 10.1007/DCR.0b013e3181bdee8c. PMID 20010354
- [Background] Hardt J, Meerpohl JJ, Metzendorf MI, Kienle P, Post S, Herrle F. Lateral pararectal versus transrectal stoma placement for prevention of parastomal herniation. Cochrane Database Syst Rev. 2019 Apr 24;4(4):CD009487. doi: 10.1002/14651858.CD009487.pub3. PMID 31016723
- [Background] Jones HG, Rees M, Aboumarzouk OM, Brown J, Cragg J, Billings P, Carter B, Chandran P. Prosthetic mesh placement for the prevention of parastomal herniation. Cochrane Database Syst Rev. 2018 Jul 20;7(7):CD008905. doi: 10.1002/14651858.CD008905.pub3. PMID 30027652